CLINICAL TRIAL: NCT06388330
Title: The Effect of a Low FODMAP Diet in Functional Dyspepsia Patients With Meal Related Symptoms (Postprandial Distress Syndrome According to the Rome IV Consensus)
Brief Title: The Effect of a Low FODMAP Diet in Functional Dyspepsia Patients With Meal Related Symptoms
Acronym: FFD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, Professor, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: s61692
Record Dates: First submitted 2020-05-06; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Functional Dyspepsia; FODMAP Diet
MeSH Terms: interventions — FODMAP Diet

STUDY DESIGN:
Masking Description: open label strict diet phase blinded participant during reintroduction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- low FODMAP diet (Experimental)
  Interventions: Other: low FODMAP diet

INTERVENTIONS:
Other: low FODMAP diet — strict low FODMAP diet followed by reintroduction of different FODMAPs and glucose (control)

SUMMARY:
In this study, the investigators will evaluate the FODMAP diet as an alternative treatment for functional dyspepsia and explore its effect on different aspects of the pathophysiology of FD.

DETAILED DESCRIPTION:
The study design starts with a baseline period of 2 weeks, includes 6 weeks of a 'strict' FODMAP diet (no blinded), followed by a 9 week 'reintroduction' phase (single blind). Based on the patients' symptom results following each of these challenges, patients will then follow the 'moderate' FODMAP diet, where the FODMAPs that did not trigger any symptoms during the challenge tests can now be consumed. Finally patients follow 2 weeks of a diet 'moderate' in FODMAP levels (no blinded). Blood and stool samples will be collected during the complete trial at several timepoints. In addition, before and after the strict diet phase a gastroscopy will be performed as well as an intragastric pressure measurement and breath test.

ELIGIBILITY:
Inclusion Criteria:

* patients with functional dyspepsia (postprandial distress syndrome)
* written informed consent
* 18-70 years

Exclusion Criteria:

1. Patients with any condition which, in the opinion of the investigator, makes the patient unsuitable for entry into the study
2. Patients with any major psychiatric disorders (including those with a major psychosomatic element to their gastrointestinal disease), depression, alcohol or substance abuse in the last 2 years
3. Patients presenting with predominant symptoms of irritable bowel syndrome (IBS) and of gastro-oesophageal reflux disease (GERD)
4. Patients who changed their diet over the last 3 months or have previously tried the low FODMAP diet are excluded from the study.
5. Females who are pregnant or lactating are excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Improvement on gastrointestinal symptoms | 2 years
  The primary endpoint is to evaluate the efficacy of low FODMAP diet on gastrointestinal symptoms in FD. Based on the LPDS questionnaire (Leuven Postprandial Distress Syndrome Score), the primary endpoint is defined. This questionnaire contains questions with a scoring system from 0 till maximum 5 with higher scores indicating higher symptom severity. An improvement of 0.5 is considered clinically meaningful.

SECONDARY OUTCOMES:
Reintroduction period | 2 years
  Percentage of patients experiencing symptom worsening upon blinded reintroduction of single FODMAPs by means of LPDS daily diaries
Evaluation of the low FODMAP diet on IBS related symptoms | 2 years
  by IBS-SSS and IBS-QoL questionnares
Evaluation of the low FODMAP diet on symptom response and quality of life | 2 years
  by PAGISYM and SFNDI questionnaires
Evaluation of the low FODMAP diet on depression, somatization | 2 years
  by PHQ
Evaluation of the low FODMAP diet on duodenal barrier function | 2 years
  Duodenal mucosal integrity was evaluated in adapted mini-Ussing chambers and defined by transepithelial electrical resistance (TEER) and paracellular permeability for FITC dextran (macromolecular flux) (4kDa).
Evaluation of the low FODMAP diet on gastric emptying | 2 years
  The C13-octanoic breath test was used to measure gastric emptying rate.
Evaluation of the low FODMAP diet on gastric accommodation | 2 years
  Intra-gastric pressure measurement was used to quantify gastric accommodation at baseline and at the end of the low FODMAP diet.

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium